CLINICAL TRIAL: NCT00000778
Title: A Pilot Study of Methodology to Rapidly Evaluate Drugs for Bactericidal Activity, Tolerance, and Pharmacokinetics in the Treatment of Pulmonary Tuberculosis Using Isoniazid and Levofloxacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: DATRI 008
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 1995-06

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Isoniazid; Tuberculosis, Pulmonary; Pyridoxine; Ofloxacin; AIDS-Related Opportunistic Infections; Drug Evaluation; Acquired Immunodeficiency Syndrome; Sputum; Colony Count, Microbial
MeSH Terms: conditions — HIV Infections; Tuberculosis; Tuberculosis, Pulmonary; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Isoniazid; Pyridoxine; Levofloxacin

INTERVENTIONS:
Drug: Isoniazid
Drug: Pyridoxine hydrochloride
Drug: Levofloxacin

SUMMARY:
To evaluate the methodology for rapidly determining the early bactericidal activity (EBA), tolerance, and pharmacokinetics of isoniazid and levofloxacin in the treatment of pulmonary tuberculosis (TB).

Traditionally, in trials for treatment of TB, a new drug is administered in combination with two or more other antituberculous agents of known effectiveness over a long period of time. In this setting, it is difficult to determine the effect of any single drug or dose level. Development of new agents for the treatment of TB may be accelerated by a methodology in which a new agent could be evaluated for activity by administering it as a single agent over a short time period. This study utilizes a method to measure the amount of bacteria present each day in the lungs.

DETAILED DESCRIPTION:
Traditionally, in trials for treatment of TB, a new drug is administered in combination with two or more other antituberculous agents of known effectiveness over a long period of time. In this setting, it is difficult to determine the effect of any single drug or dose level. Development of new agents for the treatment of TB may be accelerated by a methodology in which a new agent could be evaluated for activity by administering it as a single agent over a short time period. This study utilizes a method to measure the amount of bacteria present each day in the lungs.

An initial cohort of patients receive isoniazid (with pyridoxine) daily for 5 days. Sputum samples are collected daily for determination of the EBA (decline in colony-forming units/ml sputum). If the methodology is validated, additional patients are randomized to receive one of two doses of levofloxacin daily for 5 days, with determination of EBA. All patients are hospitalized for 2 days of baseline evaluation and 5 days of treatment.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed in all patients:

* Antacids if administered more than 2 hours before or after study drug.

Allowed in isoniazid patients:

* Anticonvulsant therapy if blood levels are monitored.

Allowed in levofloxacin patients:

* Acceptable medications other than antacids if administered at least 2 hours before or 1 hour after study drug.
* Anticonvulsant therapy, theophylline, or warfarin if doses are monitored.

Patients must have:

* Presumptive active pulmonary TB.
* No clinical evidence of central nervous system or miliary tuberculosis.

NOTE:

* Both HIV-positive and HIV-negative patients are eligible.

NOTE:

* Pregnant women may be enrolled in the isoniazid cohort only.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active or suspected MAI infection.
* Active or suspected hepatitis.
* Any other serious acute infection, diabetes, chronic obstructive pulmonary disease, malignancy requiring chemotherapy, or major organ dysfunction.
* Extreme illness or toxic appearance.
* Pregnancy (if entering the levofloxacin portion of the study).

Concurrent Medication:

Excluded:

* All standard TB therapies.
* Clofazimine.
* Rifabutin.
* Quinolones.
* Aminoglycosides.
* Corticosteroids.
* Pentoxifylline.
* Colony-stimulating factors.
* Interferons.
* Interleukins.
* Disulfiram (patients receiving isoniazid).

Patients with the following prior conditions are excluded:

* History of treatment-limiting intolerance or known hypersensitivity to isoniazid (in patients receiving isoniazid) or to quinolones (in patients receiving levofloxacin).
* Vomiting or diarrhea >= grade 2 at screening or within 2 days prior to screening.
* History of drug-resistant TB (in patients receiving isoniazid).

Prior Medication:

Excluded:

* Any prior treatment or prophylaxis for TB if enrolling on the isoniazid cohort.
* Any anti-TB drug within the past 12 weeks, including standard drugs against TB as well as clofazimine, rifabutin, and all quinolones and aminoglycosides.
* Corticosteroids, pentoxifylline, colony-stimulating factors, interferons, or interleukins within the past 12 weeks.

Known risk factors for multi-drug resistant (MDR) TB, including:

* Domicile, shelter, or prison exposure to a known case of MDR TB within the past 6 months.
* Residence in a specific domicile, shelter, or prison cell block within 6 months of a known outbreak of MDR TB.
* Hospitalization, within the past 6 months, on a medical service or unit in which nosocomial transmission of MDR TB is known to have occurred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44

CONTACTS AND LOCATIONS:
Overall Officials: Hafner R, Study Chair; Cohn J, Study Chair; Egorin M, Study Chair
Locations (10):
- United States (10):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Med Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Broward Gen Med Ctr, Fort Lauderdale, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Illinois, Chicago, Illinois
  - Tulane Univ Med School, New Orleans, Louisiana
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ TX Galveston, Galveston, Texas
  - Baylor College of Medicine / Houston Veterans Adm Med Ctr, Houston, Texas

REFERENCES:
- [Background] El-Sadr WM, Perlman DC, Matts JP, Nelson E, Cohn D, Telzak E, Chirgwin K, Salomon N, Olibrice M, Hafner R. Outcome of an induction regimen for the treatment of HIV-related tuberculosis (TB): evaluation of the addition of a quinolone. Int Conf AIDS. 1996 Jul 7-12;11(1):327 (abstract no TuB2358)